CLINICAL TRIAL: NCT05167981
Title: One-Year Impact Evaluation of Retaining Employment and Talent After Injury/Illness Network (RETAIN) in Kansas
Brief Title: RETAINWORKS Impact Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: The United States Social Security Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTN-KS
Record Dates: First submitted 2021-11-05; First posted 2021-12-22 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Disability
Keywords: disability; employment; unemployment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN Programming (Experimental): The experimental group receives the full set of RETAINWORKS intervention activities.
  Interventions: Other: RETAINWORKS
- Control (No Intervention): The control group receives information and referral to partner services.

INTERVENTIONS:
Other: RETAINWORKS — The experimental group is eligible to receive the full set of RETAINWORKS intervention activities. The program includes a combination of medical provider services, stay-at-work (SAW)/return-to-work (RTW) coordination services, and other SAW/RTW services. Participants receive intensive case management and care coordination by health and employment services RTW navigators. Financial incentives are offered to participants and medical providers for milestone attainment and training achievement.
  Arms: RETAIN Programming

SUMMARY:
The Retaining Employment and Talent after Injury/Illness Network (RETAIN) demonstration is a collaborative effort between the U.S. Department of Labor (DOL) and the Social Security Administration (SSA) to improve employment outcomes for individuals who experience injuries or illnesses that put them at risk of exiting the labor force and relying on disability programs and other public supports in the long term. RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. This evaluation will focus on the Kansas Department of Commerce's implementation of "RETAINWORKS" statewide. The evaluation will document how the project is implemented, describe enrollees, estimate the project's impacts on enrollees' outcomes, and assess whether the benefits outweigh the costs.

DETAILED DESCRIPTION:
The Kansas Department of Commerce has partnered with a consortium of medical and business partners to implement "RETAINWORKS" statewide. SSA contracted with Mathematica to conduct an independent evaluation of the program. Under the RETAIN model medical providers receive training and incentives to use occupational health best practices. The state agency also coordinates SAW/RTW services for the enrollee, fosters communication among RETAINWORKS stakeholders about the treatment enrollee returning to work, and monitors the enrollee's medical and employment progress. RETAINWORKS also uses nurse navigators and workforce coordinators to support workplace-based interventions and retain or rehabilitate enrollees. Financial incentives are offered to participants and medical providers for milestone attainment and training achievement.

Kansas recruits participants through referrals from medical providers. After initial intake by a nurse navigator, a workforce coordinator randomly assigns each enrollee to either a treatment group that is eligible to receive the full set of RETAIN intervention activities or a control group that is not. The evaluation team then compares the outcomes of the two groups and gathers evidence on how RETAINWORKS shaped the outcomes of enrollees who were eligible for its services, regardless of whether they participated in those services. Data sources include enrollment data, surveys, administrative records, program data, and qualitative data.

ELIGIBILITY:
Inclusion Criteria

* Has a work disability. Work disability is defined as an injury, illness, or medical condition that has the potential to inhibit or prevent continued employment or labor force participation. Work disability exists when an employee is not able to perform their usual work as a result of a health problem
* The work disability (i.e., illness, injury, or medical condition) must impact the participant's employment in one or more of the following ways:

  1. Participant's ability to attend work;
  2. Participant's ability to perform work duties;
  3. Participant's work performance/productivity
* The condition must be a new condition or an exacerbation of a chronic condition that falls into one or more of the following categories:

  1. Musculoskeletal injuries;
  2. Mental health disorders;
  3. Chronic diseases such as Diabetes, Chronic Obstructive Pulmonary Disease (COPD), or Congestive Heart Failure (CHF) - this list is not all-inclusive;
  4. Other newly diagnosed illnesses or injuries that affect the individual's employment
* The condition may be acquired from or attributed to either on-the-job (occupational-related) or off-the-job (non-occupational-related) factors
* The participant must meet all the following criteria:

  1. Be between the ages of 18 and 65 years;
  2. Be currently employed or seeking employment;
  3. Either live or work in Kansas;
  4. Have a valid social security number;
  5. Be legally authorized to work in the United States

Exclusion Criteria

* May NOT have application for SSDI or SSI benefits pending or already receiving such benefits at the onset of the injury or illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Share of enrollees employed in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Share of enrollees employed in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Enrollee earnings in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Sum of enrollee earnings in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Share of enrollees that applied for SSDI or SSI during the 12 months after enrollment | Measured in the 12 months after enrollment.
  Share of enrollees that applied for SSDI or SSI during any of the 12 months after enrollment obtained from SSA program data. These files include detailed information about Social Security Disability Insurance (SSDI) and Supplemental Security Income (SSI) applications SSDI and SSI awards, SSDI and SSI benefit amounts and enrollee characteristics (for enrollees who have ever applied for SSA program benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Berk, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Kansas Department of Commerce, Topeka, Kansas, United States

IPD SHARING:
Plan to Share IPD: No